CLINICAL TRIAL: NCT04480515
Title: Does COVID-19 Pandemic Reduce In-hospital Mortality?
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ramazan Guven, Professor, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KSSEAH--IHM
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Covid19; In-hospital Cardiac Arrest
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: in-hospital mortality rate — In-hospital mortality rate during pandemic of 2020 will be compared with the in-hospital mortality rate of the last year's same time period

SUMMARY:
COVID-19, which emerged in China in December 2019, has become a pandemic with its spread to many countries of the world. Although it is suggested that hospital admissions are reduced due to some reasons such as trauma, during COVID-19 pandemic, it is controversial whether in-hospital mortality rates changed. Therefore this multi-centered study aimed to determine how in-hospital mortality effected during the pandemic period according to the specific patient groups.

DETAILED DESCRIPTION:
COVID-19, which emerged in China in December 2019, has become a pandemic with its spread to many countries of the world. Although it is suggested that hospital admissions are reduced due to some reasons such as trauma, during COVID-19 pandemic, it is controversial whether in-hospital mortality rates changed. Therefore this multi-centered study aimed to determine how in-hospital mortality effected during the pandemic period according to the specific patient groups. Thus, in case of a pandemic, it will be a guide in which patient groups healthcare providers should be more careful about.

ELIGIBILITY:
Inclusion Criteria:

* Deaths, with all required data available, occurred within the study hospitals
* centers Accepted to participate with an informed consent

Exclusion Criteria:

* lack of consent
* lack of data
* deaths occurred outside the study hospitals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the records of in-hospital mortality will be evaluated
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 4 months
  During the pandemic (March-July), deaths occurred in hospital will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No